CLINICAL TRIAL: NCT06651554
Title: Harnessing Technology-assisted Methods to Advance Suicide Prevention Among Youth in Colombian School Settings
Brief Title: Technology-assisted Methods to Advance Suicide Prevention Among Youth in Colombia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00000508; R34MH136232-01 (NIH)
Record Dates: First submitted 2024-10-18; First posted 2024-10-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2024-11

CONDITIONS: Suicidal Ideations; Suicidal Behaviors; Depression, Anxiety; Well-being
Keywords: suicide prevention; adolescent health; mHealth; Colombia; Implementation Science
MeSH Terms: conditions — Suicidal Ideation; Depression; Anxiety Disorders; Suicide Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital Platform Intervention (Experimental): Key features of the digital platform intervention include mental health self-help tools, a customizable safety plan, links to online counseling services, and gamification elements.
  Interventions: Behavioral: Digital Platform Intervention
- waitlist control (No Intervention): No intervention will be administered to youth during their assigned waitlist control period.

INTERVENTIONS:
Behavioral: Digital Platform Intervention — Key features of the digital platform include mental health self-help tools, a customizable safety plan, links to online counseling services, and gamification elements. Youth will be able to access the digital platform as often as they like during their assigned 3-month intervention period.
  Arms: Digital Platform Intervention

SUMMARY:
This study will investigate a multi-level approach that applies technology-assisted methods to reduce suicidal thoughts and behaviors (SIB) and promote mental health among Colombian youth: (a) digital platform for youth; (b) digital platform for teachers; and (c) hybrid mental health training diploma program for teachers. This approach will evaluate an open-access digital platform for suicide prevention among Colombian youth. Key features of the digital platform include mental health self-help tools, a customizable safety plan, links to online counseling services, and gamification elements. The digital platform's teacher interface will incorporate psychoeducation, brief suicide-risk screening and decision support tools to enhance teacher capacity to assess risk for suicide and refer youth to the appropriate level of services.

Study investigators will conduct a hybrid-type 1 implementation-effectiveness stepped wedge pilot trial design to evaluate the digital platform and hybrid mental health teacher training program implemented within secondary schools in Bogota, Colombia. Study aims are to:

Aim 1. An initial needs assessment will be conducted with key stakeholders (youth, teachers, caregivers, school administrators) to identify barriers and facilitators to successful implementation of the multi-level approach. User-centered design methods will be used to refine the digital platform and incorporate end-user feedback into the final prototype.

Aim 2. Investigators will evaluate: (a) feasibility, acceptability, and usability of the digital platform across three schools in Colombia; and (b) the preliminary effects of the digital platform in reducing SIB and improving mood (e.g., anxiety/depression) among Colombian youth aged 14-19 attending the three schools. Safety planning skills acquisition (youth-level) and linkages to mental health services (service-level) will be assessed as potential mechanisms of change.

Aim 3. The study will apply a multi-disciplinary capacity building model to strengthen behavioral health and implementation science research, healthcare delivery capacity, and mental health policy. In partnership with Pontificia Javeriana University, experts in suicide prevention, data science, and implementation science will be engaged to build in-country research capacity at the individual and institutional level.

DETAILED DESCRIPTION:
This study uses a multi-level approach that leverages innovative, culturally appropriate mHealth technology to reduce SIB and promote mental health in Colombian youth: (a) digital platform for youth; (b) digital platform for teachers; and (c) hybrid mental health training program for teachers. Study investigators will conduct a hybrid-type 1 implementation-effectiveness stepped wedge pilot trial to evaluate the digital platform and hybrid mental health teacher training program implemented within secondary schools in Bogota, Colombia.

Prior to launching the pilot trial, study investigators will conduct an initial needs assessment with key stakeholders to identify barriers and facilitators to successful implementation of the digital platform. Investigators will use a mixed methods approach and conduct qualitative interviews with key stakeholders (teachers (N=10), youth (N=12), caregivers (N=5) and school administrators (N=3)). Quantitative measures will include school climate, leadership, and attitudes towards technology-assisted interventions. Qualitative data analysis will follow an iterative process of open coding for themes, followed by focused coding to determine frequency of themes. Mixed methods analysis will use joint displays to integrate qualitative and quantitative data and highlight key findings. Results will inform development of a formal implementation blueprint that will be reviewed with key stakeholders and used to guide implementation of the platform.

User-centered design methods will guide refinements of the youth interface and further development of the teacher interface in the digital platform. The process will include two co-design workshops with youth (N=10) and two with teachers (N=8). Ender-user feedback from the initial co-design process will be incorporated to further optimize the digital platform's functionality and features to build the alpha prototype. Three, iterative user-testing sessions of the alpha prototype will be held with youth and teachers using "think aloud protocols" to elicit end-user feedback on features that are user-friendly versus confusing or hard to use. Feedback from user-testing sessions will inform further refinements and development of the beta prototype. Study investigators will then conduct three additional user-testing sessions with teachers and youth, respectively, to test the beta prototype. User-testing participants will complete the System Usability Scale after the last UI/UX testing session to asses usability prior to launching the pilot trial.

Aim 1. (Exploration and Preparation) Explore barriers and facilitators to successful implementation of the digital platform in Colombian schools. A mixed-methods participatory process with key stakeholders will be used to identify implementation barriers and facilitators. Aim 1a. User-centered design principles will guide refinements of the digital platform.

Aim 2. (Implementation) Conduct a hybrid type 1 implementation-effectiveness stepped wedge pilot trial to assess the feasibility, acceptability, usability and preliminary effects of the digital platform implemented within 3 schools in reducing SIB and improving mood (e.g., anxiety/depression) among Colombian youth aged 14-19 (N=150). Study Hypotheses are that: (a) the digital platform will be feasible, acceptable, and usable among youth; and (b) youth who use the digital platform will exhibit greater reductions in SIB and mood symptoms during their school's intervention period compared with youth in the pre-intervention period (no digital platform use) at post-intervention and 3-month follow-up. Aim 2a. Explore safety planning skills (youth-level) and linkages to mental health services (service-level) as mechanisms of change. We hypothesize that: (a) use of the digital platform will be related to greater safety planning skills and service usage; and (b) safety planning skills and service usage will be related to reduced SIB and mood symptoms.

Study investigators will conduct a hybrid type 1 implementation-effectiveness stepped wedge pilot trial to evaluate digital platform implementation in Colombian schools. A hybrid type 1 implementation-effectiveness design, even if it is only a pilot study, will support the evaluation of SIB and mood symptoms as primary outcomes, with implementation outcomes as secondary. Because there are signficant ethical and logistical issues posed by randomizing schools to a study condition, a stepped wedge design is a pragmatic option that will allow for sequential transition of each school to the intervention condition in a randomized order. The stepped wedge design has been used successfully in prior studies of school-based interventions in LMICs. A complete stepped wedge design measures outcomes from all clusters (e.g., schools) at every data collection time point, regardless of intervention exposure; however, due to resource and time constraints, this study will use an incomplete stepped wedge design in which study outcomes are measured at three timepoints for each school.

The research team will recruit and enroll three secondary schools in Bogota to participate in the hybrid type 1 pilot stepped wedge trial. Selection guidelines for schools will also include rules to minimize risk of contamination (i.e., geographical distance between schools). Enrolled schools will be randomized to a sequence, which includes time exposed to the digital platform and mental health training program for teachers. Intervention exposure periods will be 3-months in duration, which will provide sufficient time for teachers to complete the hybrid mental health training program and for youth to access and use the digital platform as needed. The research team will then recruit and enroll youth (N=228; 76 per school) and teachers (N=30; 10 per school) from enrolled schools, with stratified selection to aim for gender balance in recruitment. Youth and teachers will complete quantitative assessments during their school's baseline, post-intervention, and 3-month follow-up period.

Digital platform implementation with youth and teachers: there will be one initial in-person, 1-hr introductory session with enrolled youth and one with teachers to provide an overview of the digital platform's features and functions. Youth and teachers will have the opportunity to test out the digital platform and ask questions. After the introductory session, youth and teachers will be able to create an account to access the digital platform and use the different available tools as often as they choose, at the time they choose, during the 3-month intervention period. Digital platform data will be stored in a HIPAA compliant could-based storage system and backed up on a HIPAA compliant server at Javeriana University. All data will be deidentified to protect personal privacy and confidentiality of participants. Technical assistance will be available to address any bugs or technology challenges encountered by participants.

Central features of the digital platform include: (a) integration with social media for easy youth access; (b) authentication and guardian consent; (c) mental health screening; (d) linkages with online mental health counseling; (e) customizable safety planning; and (f) gamification elements. The platform also includes self-help tools incorporating key components of evidence-based mental health interventions with a transdiagnostic focus (i.e., cognitive-behavioral therapy, mindfulness-based approaches) that have shown effectiveness in reducing symptoms across a range of mental health disorders.

Hybrid mental health teacher training program implemention: Our certified teacher training program consists of 120 didactic hours across a 3-month period. It includes six modules: (1) Introduction to mental health and academic performance; (2) Addressing emotions in childhood and adolescence; (3) Substance use (legal and illegal) in children and adolescents and eating behavior; (4) Aggressive behaviors and bullying in schools; (5) Sexuality, suspected sexual abuse, and mistreatment; (6) Inclusive education and resilience. The second module contains evidence-based tools for identifying suicide risk and warning signs as well as to guide referrals for psychiatric emergency assessment and/or other services. The training program is completed with synchronous sessions as well as asychronous participation. The duration of each module is about 2 weeks.

Primary Outcomes will be measured via quantitative assessments at the youth participant level and include SIB, depression, anxiety, well-being, and safety planning skills. Secondary Outcomes will be assessed at both the youth and teacher level and include feasibility, acceptability, usability and appropriateness of the digital platform via qualitative interviews conducted at post-intervention. Teacher participant level mental health literacy, sense of self-efficacy, and satisfaction with the hybrid mental health training program will also be assessed via quantitative assessments. All quantitative assessments will be administered at baseline, post-intervention, and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria for youth:

* aged 14-19
* attending a secondary school in Bogota
* willing to try the digital platform

Exclusion Criteria for youth:

* not meeting inclusion criteria

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 | Baseline, immediately after the intervention, and 3-months after the intervention
  The PHQ-9 is a 9-item scale used as a brief assessment of depression symptoms during the past two weeks. The measure is scored on a 4-point Likert scale: 0=not at all; 1=several days; 2=more than half the days; 3=nearly every day. Higher scores indicate worse depression symptoms. Item 9 can be used to screen for suicidal ideation (e.g., thoughts that you would be better of dead or hurting yourself). The measure has been translated to Spanish and validated previously in Colombia with youth and adults.
GAD-7 | baseline, immediately after the intervention and 3-months after the intervention
  The GAD-7 is a 7-item scale used as a brief assessment of anxiety symptoms. The measure is scored on a 4-point Likert scale: 0=not at all; 1=several days; 2=more than half the days; 3=nearly every day. Higher scores indicate worse anxiety. The measure has been translated to Spanish and validated previously in Colombia with youth and adults.
Self-injurious Thoughts and Behaviors Interview-short form, adapted | baseline, immediately after the intervention and 3-months after the intervention
  The SITBI short form is a structured interview designed to assess the presence, frequency, and characteristics of a broad array of self-injurious thoughts and behaviors. The measure has been translated to Spanish and validated in adolescent/young adult and Spanish speaking populations. Items are scored on a 5-point Likert-scale ranging from: 0=low/little to 4=very much/severe. Higher scores indicate greater frequency and/or severity of self-injurious thoughts and behaviors.

SECONDARY OUTCOMES:
WHO-5 | baseline, immediately after the intervention and 3-months after the intervention
  The WHO-5 is a 5-item scale that measures current well-being over the past two weeks. The measure is scored on a 6-point Likert-scale: 0=at no time; 1=some of the time; 2=less than half of the time; 4=most of the time; 5=all of the time. Higher scores reflect a greater sense of well-being. The measure has been translated to Spanish and validated with populations of youth and adults.

CONTACTS AND LOCATIONS:
Overall Officials: Alethea Desrosiers, Principal Investigator — Brown University
Locations (1):
- Pontificia Javeriana Universidad, Bogotá, Colombia, Colombia

IPD SHARING:
Plan to Share IPD: No
The study team does not plan to publish in the ICMJE journals.